CLINICAL TRIAL: NCT00493038
Title: Prospective, Multicenter, Randomized, Double Blind, Parallel Arm Study to Evaluate the Efficacy and Safety of Moxifloxacin 400 mg OD for 7 Days Versus a Standard Antibiotic Therapy for 10 Days in the Treatment of Acute Bacterial Rhino Sinusitis
Brief Title: Study to Evaluate the Efficacy and Safety of Moxifloxacin Versus Amoxicillin/Clavulanate in the Treatment of Acute Bacterial Rhinosinusitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was prematurely terminated due to slow enrollment beyond the planned study timelines.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11881; 2005-002779-34 (EudraCT Number)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2009-04-13 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Sinusitis; Bacterial Infections
Keywords: Treatment of acute bacterial rhinosinusitis
MeSH Terms: conditions — Sinusitis; Bacterial Infections | interventions — Moxifloxacin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Avelox, BAY12-8039) (Experimental): Moxifloxacin (Avelox, BAY12-8039) 400 mg tablets once daily (OD) for 7 days and amoxicillin/clavulanate 1000 mg matching placebo tablets three times daily (TID)for 10 days
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Amoxicillin/Clavulanate (Active Comparator): Amoxicillin/clavulanate 1000 mg tablets three times daily (TID) for 10 days and moxifloxacin 400 mg matching placebo tablets once daily (OD) for 7 days
  Interventions: Drug: Amoxicillin/Clavulanate

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Patients will be administered daily a single moxifloxacin 400 mg tablet for 7 days
  Arms: Moxifloxacin (Avelox, BAY12-8039)
Drug: Amoxicillin/Clavulanate — Patient will be administered daily Amoxicilline/Clavulanate 1000 mg tablets every 8 hours for 10 days
  Arms: Amoxicillin/Clavulanate

SUMMARY:
This is a clinical study organized to collect clinical data to better define the activity of some antimicrobials already marketed in Italy and in the rest of the world for the treatment of acute bacterial rhinosinusitis

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Clinical diagnosis of acute rhinosinusitis with signs and symptoms present for >/= 5-7 days but < 28 days
* Clinical diagnosis will be confirmed by nasal endoscopic examination

Exclusion Criteria:

* History of chronic sinusitis defined as greater than four weeks of continuous symptoms (subject with history of sinus surgery may be included; subjects with recurrent acute sinusitis may be included)
* Any symptoms that suggest the subject's current illness is allergic rhinitis (e.g. repetitive sneezing, itchy nose or eyes, provocation by an allergen) and not acute bacterial sinusitis
* Known bacteremia, meningitis or infection infiltrating the tissues neighboring the sinuses
* Known immunodeficiency diseases including, but not limited to: neutropenia (neutrophil count < 1000/mm3), human immunodeficiency virus (HIV) infection (Cluster of differentiation 4 (CD4)+ T-cell count of < 200/mm3). Note: HIV testing is not required
* Received systemic antibacterial therapy likely to be effective in the treatment of acute bacterial sinusitis for more than 24 hours within 5/6 days of enrollment
* Requirement for concomitant systemic antibacterial therapy with agents other than those specified in this protocol
* Currently receiving topical nasal corticosteroids, unless they have been on a stable dose for > 4 weeks prior to enrollment
* Requirement for concomitant therapy with systemic corticosteroids
* Pregnant or breast feeding
* Of childbearing potential in whom pregnancy cannot be excluded by a negative pregnancy test and who are not using reliable barrier method of contraception
* Received an investigational drug in the past 30 days
* Previously enrolled in this study
* Unable to take oral medication
* History of allergy to quinolone antibiotics or related compounds and beta-lactams
* History of tendinopathy associated with quinolones
* Known to have congenital or sporadic syndromes of QT interval corrected for rate (QTc) prolongation or receiving concomitant medication reported to increase the QTc interval (e.g. amiodarone, sotalol, disopyramide, quinidine, procainamide, terfenadine)
* Uncorrected hypokalemia
* End stage liver cirrhosis (class Child-Pugh C)
* Severe renal impairment requiring dialysis
* Diagnosis of rapidly fatal illness with a life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- Italy (29):
  - San Benedetto del Tronto, Ascoli Piceno
  - Esine, Brescia
  - Lamezia Terme, Catanzaro
  - Cesena, Forlì
  - Sestri Ponente, Genova
  - Monza, Monza-Brianza
  - Comiso, Ragusa
  - Bari
  - Benevento
  - Bergamo
  - Bologna
  - Bolzano
  - Caserta
  - Catania
  - Florence
  - Foggia
  - Lecce
  - Lecco
  - Matera
  - Milan
  - Novara
  - Pavia
  - Perugia
  - Pisa
  - Roma
  - Siena
  - Torino
  - Treviso
  - Udine

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started on 13 Feb 2006 and the last study visit occurred on 20 Jan 2008. The study was conducted at 34 active otorhinolaryngology centers in Italy.
Pre-assignment Details: Number of patients screened: 293 Number of patients having at least one observation under study medication: 287 (intention-to-treat population = ITT population) Number of patients adhered to major predefined aspects of the study protocol: 251 (per-protocol population = PP population). Primary population for efficacy was PP.
Groups:
- Moxifloxacin (Avelox, BAY12-8039): Moxifloxacin (Avelox, BAY12-8039) 400 mg tablets once daily (OD) for 7 days and amoxicillin/clavulanate 1000 mg matching placebo tablets three times daily (TID) for 10 days
- Amoxicillin/Clavulanate: Amoxicillin/clavulanate 1000 mg matching tablets three times daily (TID) for 10 days and moxifloxacin 400 mg matching placebo tablets once daily (OD) for 7 days
Period: Treatment
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Started | 147 | 146
Randomization | 147 | 146
Treated With Study Medication | 145 | 142
Test-of-Cure Visit | 123 | 126
Completed | 123 | 126
Not Completed | 24 | 20
Not completed — Adverse Event | 8 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Other | 0 | 1
Period: Follow-up
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Started | 123 | 126
Completed | 122 | 126
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate | Total
Number analyzed (Participants) | 145 | 142 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13.2) | 39.7 (13.6) | 40.7 (13.4)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  >18 and <65 years | 133 | 132 | 265
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 75 | 138
  Male | 82 | 67 | 149

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response (Per-protocol Population)
Description: Number of patients in the population who met criteria pre-specified in the protocol whose clinical response 1-3 days after treatment was assessed by the investigator as "clinical cure"
Time Frame: At 'Test-of-Cure', Day 1-3 after treatment
Population: Per Protocol population: subjects to meet all of the following (1) Clinical evaluation was performed at TOC visit (2) No other systemic antibacterial agent was administered with study drug up to TOC visit (3) Adequate treatment compliance (≥ 80% of study drug taken) (4) Random code not broken (5) No protocol violation affecting treatment efficacy
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Number analyzed (Participants) | 121 | 130
participants | 119 | 125
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Amoxicillin/Clavulanate; Calculated were 95% confidence intervals for the difference in success rates between treatment groups (moxifloxacin minus comparator). Method as described in Koch et al. ('Categorical Data Analysis' in Statistical methodology in the pharmaceutical sciences / edited by D. A. Berry, p. 415 ff., Marcel Dekker, 1990); Test type: Non-Inferiority or Equivalence — The non-inferiority margin was set to 15% in the protocol. Sample size was estimated using the method as described in Farrington-Manning (STATISTICS IN MEDICINE, Vol. 9; Farrington CP, Manning G: "Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference...", pg.1447-1454 [1990]). Estimation was performed to achieve 90% power, based on the equivalence delta of 15%, and a clinical success rate of 80% in the per protocol population; Mean Difference (Final Values) = 2.1, 95% CI [-1.9 to 6.2] — Mean difference denotes the difference of clinical cure rates between the two treatment groups (moxifloxacin minus amoxicillin/clavulanate)

2. Secondary Outcome: Number of Participants With Response (Intent-to-treat Population)
Description: Number of patients in the population who received at least one dose of study medication whose clinical response 1-3 days after treatment was assessed by the investigator as "clinical cure"
Time Frame: At 'Test-of-Cure', Day 1-3 after treatment
Population: ITT population: participants having at least one observation under study medication
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Number analyzed (Participants) | 145 | 142
participants | 128 | 127
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Amoxicillin/Clavulanate; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI [-7.9 to 6.8]

3. Secondary Outcome: Number of Participants With Response (Per-protocol Population)
Description: Number of patients in the population who met criteria pre-specified in the protocol whose clinical response 24-30 days after treatment was assessed by the investigator as "continued clinical cure"
Time Frame: End of Follow-up, Day 24-30 after treatment
Population: PP population at end FU: (1) Clinical evaluation was performed at the TOC visit (2) No other systemic antibacterial agent was administered with study drug up to the TOC visit (3) Adequate treatment compliance (≥80% of study drug taken) (4) Random code not broken (5) No protocol violation affecting treatment efficacy (6) FU assessment available
Measure: Number; unit: participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Number analyzed (Participants) | 113 | 124
participants | 108 | 117
Statistical Analysis 1: Comparison: Moxifloxacin (Avelox, BAY12-8039) vs Amoxicillin/Clavulanate; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.7, 95% CI [-3.8 to 7.1]

4. Secondary Outcome: Number of Participants With Response (Microbiologically Valid Patients)
Description: Bacteriological Efficacy Rate at the 'Test-of-Cure' visit, measured in patients defined as 'microbiologically valid'. A bacteriological success is an eradication without super- or reinfection or presumed eradication.
Time Frame: At 'Test-of-Cure', Day 1-3 after treatment
Population: Patients valid per protocol with a causative organism cultured.
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Number analyzed (Participants) | 21 | 26
Participants
  Bacteriological success | 21 | 25
  Failure | 0 | 1

5. Secondary Outcome: Number of Participants With Response (Microbiologically Valid Patients)
Description: Bacteriological Efficacy Rate at the End of Follow-up period, measured in patients defined as 'microbiologically valid'. A bacteriological success is an eradication without super- or reinfection or presumed eradication.
Time Frame: End of Follow-up, Day 24-30 after treatment
Population: Patients valid per protocol with a causative organism cultured.
Measure: Number; unit: Participants
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Number analyzed (Participants) | 21 | 26
Participants
  Bacteriological success | 19 | 23
  Failure | 0 | 0
  Missing / Indeterminate | 2 | 3

ADVERSE EVENTS:
Arm/Group | Moxifloxacin (Avelox, BAY12-8039) | Amoxicillin/Clavulanate
Serious Adverse Events (participants affected / at risk) | 1/145 | 1/142
Other Adverse Events (participants affected / at risk) | 0/145 | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (Avelox, BAY12-8039) (N=145) | Amoxicillin/Clavulanate (N=142)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to slow enrollment beyond the planned study timelines.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the trial as well as any discoveries and inventions, are exclusive property of the Promoter.

Publications on scientific review, comments or presentations about the study in scientific environment must be agreed between the Sponsor and the investigator who engages to submit to Bayer, any publication by sending one text or presentations at least 60 days before the expected publication for comments and corrections.